CLINICAL TRIAL: NCT03342183
Title: Reducing Hemodialysis Induced Recurrent Brain Injury to Improve Patients' Lives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Director of Kidney Clinical Research Unit, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109413
Record Dates: First submitted 2017-10-16; First posted 2017-11-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Disease
Keywords: Dialysis; Hemodialysis; Remote Ischemic Preconditioning
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): RIPC stimulus will be applied prior to the first intervention visit, using a previously validated (for cardiac protection in HD patients) standard dose (four cycles of cuff inflation to the lower limb of the patient and inflating at 200mmHg for five minutes, with five minutes' deflation). To be administered on a monthly basis from the baseline visit to the year 1 visit.
  Interventions: Other: Intervention Arm
- Control Arm (Sham Comparator): Sham procedure in which the blood pressure cuff will be applied to the lower limb and inflated to 40mmHg for five minutes and deflated for five minutes with the cycle repeated a total of four times prior to dialysis. To be administered on a monthly basis from the baseline visit to the year 1 visit.
  Interventions: Other: Control Arm

INTERVENTIONS:
Other: Intervention Arm — RIPC stimulus will be applied prior to the first intervention visit, using a previously validated (for cardiac protection in HD patients) standard dose (four cycles of cuff inflation to the lower limb of the patient and inflating at 200mmHg for five minutes, with five minutes' deflation).
  Arms: Intervention Arm
Other: Control Arm — Sham procedure in which the blood pressure cuff will be applied to the lower limb and inflated to 40mmHg for five minutes and deflated for five minutes with the cycle repeated a total of four times prior to dialysis. To be administered on a monthly basis from the baseline visit to the year 1 visit.
  Arms: Control Arm

SUMMARY:
Patients who receive dialysis for kidney failure suffer severe cognitive impairment. Hemodialysis causes circulatory stress and ischemia, which causes severe brain injury. It has been demonstrated that a procedure known as Remote Ischemic Preconditioning(RIPC), which involves wrapping a blood pressure cuff around a patient's leg and inflating has the potential of protecting many organs, such as the heart from the effects of dialysis. Our study aims to investigate this phenomenon to determine the extent to which it provides protection to a dialysis patient's brain.

DETAILED DESCRIPTION:
Hemodialysis patients suffer severe cognitive impairment: Abnormalities of cognitive impairment (predominately sub-cortical defects in executive decision making) are almost universal in hemodialysis (HD) patients and appear early after starting dialysis. Around 75% of patients exhibit mild cognitive impairment (MCI) and a high proportion (˜15%) have dementia. Mechanisms of injury: It has been demonstrated that HD associated circulatory stress and recurrent regional ischemia drives brain injury. The extent of injury is determined by the degree of BP instability during HD. Peritoneal dialysis patients are not subject to the same stress and retain cognitive abilities. The injury is multifactorial, and amenable to HD based intervention. Optimizing dialysis to minimize harm requires understanding the wide range of potential of pathophysiological processes contributing to this injury. Putative components of pathophysiology that might be amenable to intervention include: a) Direct reduction in tissue perfusion is the characteristic consequence of HD driven multi-organ injury. The investigators have directly visualized this in multiple organ beds during dialysis (heart, gut and kidney), and have inferred it in the brain from the development of ischemic based white matter (WM) injury. b) Inflammation drives WM injury.Endotoxin (derived from gut bacteria) is profoundly pro- inflammatory and translocates from intestinal lumen into the circulation during HD treatment directly causing WM inflammation. Daily HD (gentler fluid removal) normalizes endotoxemia and markers of inflammation. c) Release of the excitotoxic neurotransmitter, glutamate, produces injury in ischemia. Plasma levels are lower in HD patients with less ongoing brain injury. Removal of glutamate by dialysis significantly reduces ischemic injury severity and functional consequences. Previous success in protecting the brain during dialysis: The Investigator recently completed a successful multi- centre RCT of cooled dialysis fluid to abrogate WM progressive injury- strongly supporting the integral role that the HD process plays in brain injury. Hemodialysis patients have specific patterns of progressive brain injury: Currently the problem of dialysis induced functionally significant brain injury is typically not well recognized or a focus of care. Leukoaraiosis describes rarefaction of brain WM, typically associated with vascular cognitive impairment. It is universally present in HD patients (even when correcting for BP). Severity of reduction in cognitive function is proportional to the amount of WM injury, with a predominant loss of subcortical functions (executive functioning). The Investigators have previously demonstrated that the signature of the change in fractional anisotropy in dialysis patients was entirely explained by changes in radial diffusivity, rather than axial diffusivity- pathognomonic of a vascular etiology. Urgent need to develop additional interventions: Although dialysis fluid cooling appears to be effective in helping to protect against WM injury, there are limitations. The degree of cooling that can be applied is limited in some patients by cold symptom tolerability and effectiveness has only been tested in patients new to HD. Patients with more established injury may require additional therapies. These need to be suitable for combination with other emerging dialysis based therapies. Ideally they will be universally applicable, independent of dialysis machine type, low-cost, safe, well tolerated, and simple-requiring few healthcare resources to apply. Remote ischemic preconditioning (RIPC): Ischemic conditioning occurs when a transient non-lethal episode of ischemia reduces the effect of a subsequent larger insult. Similar levels of protection can be achieved by applying brief episodes of ischemia (with a BP cuff on a limb) remote from a target organ. Successful clinical studies using RIPC have been performed to provide protection against ischemia in many organs, including acute stroke, and can prevent leukoaraiosis in animal models. RIPC provides protection against HD-induced acute myocardial injury: The investigators have recently completed a pilot RCT demonstrating a RIPC intervention reduced HD-induced acute cardiac injury by 50%, after only a single application. This effect was maintained over a period of 28 days. RIPC was effective, safe and well tolerated. The investigators are currently engaged in a larger Canadian based study to refine the optimum RIPC regime to provide protection against HD-induced cardiac injury. Interim analysis of this study has confirmed similar levels of efficacy in a Canadian population and allowed us to select the maximally effective RIPC regime, for use in the current proposed study. Clear translational pathway: This project is conceived in an integrated framework of new therapeutic target discovery, intervention development and sequential testing of safety and efficacy. The investigators will use clinically relevant surrogate imaging endpoints for rapid evaluation and refinement of candidate intervention, prior to large-scale testing with survival-based endpoints. The Investigators have already developed a prototype phase III equivalent study. MY-TEMP is an Ontario based cluster randomized study of individualized dialysate cooling (trials registration NCT 02628366), funded in partnership by the Heart and Stroke Foundation, Ontario Ministry of Health and US based large dialysis provider organizations. All 7000 patients will be randomized in Q3 2016. Impact: HD patients characteristically suffer from cognitive impairment. Understanding the mechanisms behind this will allow the development of therapies integrated into dialysis treatment delivery (anti-ischemic, but potentially also directed at issues such as inflammation and dialyzable injury factors), helping patients maintain cognitive vitality, independence and maximize quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Having hemodialysis treatment at least three times per week
* Must be 18 years old or older.
* Ability to speak and understand English

Exclusion Criteria:

* Exposure to hemodialysis for less than 90 days prior to recruitment
* Established severe cognitive impairment (Montreal Cognitive Assessment test (MoCA) of less than 18 or with a formal diagnosis of dementia)
* Previous clinical stroke
* Taking drugs to blunt response to RIPC (e.g. ciclosporin, ATP-sensitive potassium channel directed drugs)
* Dialysing using lower limb vascular access
* Pregnancy, breastfeeding, or intending pregnancy
* Unable to give consent or understand written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Neuro-protection against functionally significant new brain injury | 1 year
  Change from baseline in brain damage as observed by progressive ultrastructural white matter changes on MRI imaging.

SECONDARY OUTCOMES:
Brain Perfusion | 1 year
  Change of brain perfusion from baseline MRI.
Excitotoxic neurotransmitter release | 1 year
  Change in Exitotoxic neurotransmitter release from baseline as seen on the combined MRI.
Microglial Inflammation | 1 year
  Change in microglial Inflammation from baseline as seen on the combined MRI.
Neurological impact | 1 year
  Compare observed brain injury, as determined by MRI, to results on neurocognitive test.
Depression scoring | 1 year
  Compare observed brain injury, as determined by MRI, to results on depression scoring test.We will be utilizing the PHQ-9(Patient Health Questionnaire) which is used for screening, diagnosing, monitoring, and measuring the severity of depression. This test consists of 9 questions regarding symptoms which factor into the scoring severity index. Each question is given a score from 0-3, which represents responses such as: not at all(0), several days(1), more than half the days (2), and nearly everyday(3). The scores can be interpreted as follows: 5-9 (minimal symptoms), 10-14 (Minor depression, mild), 15-19 (major depression, moderately severe), and >20 (major depression, severe).
Daily activities | 1 year
  Compare observed brain injury, as determined by MRI, to results on evaluation of activities of daily living survey.
Blood work- blood count | 1 year
  1 year results will be compared to baseline.
Blood work-urea | 1 year
  1 year results will be compared to baseline.
Blood work-microparticles | 1 year
  1 year results will be compared to baseline.
Blood work-Cardiac biomarkers (Troponin T, nTproBNP) | 1 year
  1 year results will be compared to baseline.
Blood work-CRP (C-Reactive Protein) | 1 year
  1 year results will be compared to baseline.
Blood work-glucose | 1 year
  1 year results will be compared to baseline.
Blood work- lactate | 1 year
  1 year results will be compared to baseline.
Blood work- electrolytes | 1 year
  1 year results will be compared to baseline.
Echocardiogram | 1 year
  Correlated to brain perfusion as well as circulatory stress outputs obtained by the CVInsight devices.
CVInsight | 1 year
  Help us to understand if the CVInsight® Patient Monitoring & Informatics System can be a predictor of organ perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McIntyre, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Anazodo UC, Wong DY, Theberge J, Dacey M, Gomes J, Penny JD, van Ginkel M, Poirier SE, McIntyre CW. Hemodialysis-Related Acute Brain Injury Demonstrated by Application of Intradialytic Magnetic Resonance Imaging and Spectroscopy. J Am Soc Nephrol. 2023 Jun 1;34(6):1090-1104. doi: 10.1681/ASN.0000000000000105. Epub 2023 Mar 9. PMID 36890644